CLINICAL TRIAL: NCT00604500
Title: An Open-Label, Multi-Center, Patient Handling Study of Mometasone Furoate/Formoterol Fumarate MDI With an Integrated Dose Counter in Adolescent and Adult Subjects and Adult With Asthma or COPD
Brief Title: A Patient Handling Study of Mometasone Furoate/Formortoral Fumarate (MF/F) Metered Dose Inhaler (MDI) With an Integrated Dose Counter in Adolescent and Adult Subjects With Asthma or Chronic Obstructive Pulmonary Disease (Study P04703AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04703; 3462123
Record Dates: First submitted 2008-01-21; First posted 2008-01-30 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MF/F MDI 100/10 mcg BID with dose counter (Experimental): MF/F MDI 100/10 mcg BID with an integrated dose counter (administered as two inhalations of MFF MDI 50/5 mcg, twice a day) over a 4-week Treatment Period.
  Interventions: Drug: SCH No. 418131 (Mometasone Furoate/Formoterol Furoate abbreviated MF/F )

INTERVENTIONS:
Drug: SCH No. 418131 (Mometasone Furoate/Formoterol Furoate abbreviated MF/F ) — MF/F MDI 100/10 mcg BID with an integrated dose counter (administered as two inhalations of MF/F MDI 50/5 mcg, twice a day) over a 4-week Treatment Period.

SUMMARY:
This was an open-label, multiple-dose, study of mometasone furoate/formoterol fumarate (MF/F) metered dose inhaler (MDI) 100/10 micrograms (mcg) twice daily (BID) (2 puffs of MF/F MDI 50/5 mcg, administered twice a day approximately 12 hours apart) in participants 12 years of age or older, with a diagnosis of persistent asthma or chronic obstructive pulmonary disease (COPD) of at least 12 months. The primary purpose of the study was to evaluate the performance of the MF/F MDI integrated dose counter under normal patient handling conditions.

ELIGIBILITY:
Diagnosis and Criteria for Inclusion:

* A participant must have been at least 12 years of age, of either sex, and of any race, with a diagnosis of persistent asthma or COPD of at least 12 months.
* A participant must have been able to demonstrate correct use of an MDI without a counter at the Screening Visit.
* A participant must have demonstrated at least 90% compliance with completion of the e-diary, use of the counterstrip, and use of the study medication over the 2-week Screening Period.

Exclusion Criteria:

* Participants with a serious uncontrolled medical disorder, which in the judgment of the investigator, could have interfered with the study, or required treatment which might interfere with the study.
* Participants who in the judgment of the investigator and/or sponsor had a significant recent or current, repetitive strain injury (RSI) that may have impacted their ability to effectively participate in the full duration of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2008-11-01 (Actual); Study Completion 2008-11-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weinstein C, Staudinger H, Scott I, Amar NJ, LaForce C. Dose counter performance of mometasone furoate/formoterol inhalers in subjects with asthma or COPD. Respir Med. 2011 Jul;105(7):979-88. doi: 10.1016/j.rmed.2011.01.013. Epub 2011 Mar 12. PMID 21398104

RESULTS

PARTICIPANT FLOW:
Groups:
- MF/F MDI 100/10 mcg BID (With Dose Counter): MF/F MDI 100/10 mcg BID with an integrated dose counter (administered as two inhalations of 50/5 mcg, twice a day) over a 4-week Treatment Period.
Period: Overall Study
Arm/Group | MF/F MDI 100/10 mcg BID (With Dose Counter)
Started | 272
Completed | 261 (There were 233 participants who took at least 90% of the labeled actuations (Completer Population).)
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 2
Not completed — Treatment Failure | 1
Not completed — Withdrawal by Subject | 4
Not completed — Administrative | 1
Not completed — Did not meet protocol eligibility | 1

BASELINE CHARACTERISTICS:
Arm/Group | MF/F MDI 100/10 mcg BID (With Dose Counter)
Number analyzed (Participants) | 272
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age 12 to <18 years of age | 14.69 (1.64)
  Age 18 to <65 years of age | 44.22 (12.12)
  Age ≥ 65 years of age | 70.43 (4.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 94
Number of Participants with Asthma and Chronic Obstructive Pulmonary Disease (COPD) [Number; unit: Participants]
  Asthma | 222
  Chronic Obstructive Pulmonary Disease (COPD) | 50

OUTCOME MEASURES:

1. Primary Outcome: Overall Discrepancy Rate
Description: Overall discrepancies refer to the difference between the participant-recorded number of actuations and the participant-recorded dose counter readout across the 4-week Treatment Period. The Overall Discrepancy Rate was calculated as 100 multiplied by the total number of discrepancies across all participants who used at least 90% of the labeled actuations divided by the total number of actuations in the same participant population (Completer Population).
Time Frame: 4-week Treatment Period
Population: Completer population, defined as participants who recorded use of at least 90% of the labeled actuations during the 4-week Treatment Period.
Measure: Number; unit: Overall discrepancies per 100 actuations
Arm/Group | MF/F MDI 100/10 mcg BID (With Dose Counter)
Number analyzed (Participants) | 233
Overall discrepancies per 100 actuations | 0.13

2. Primary Outcome: Overall Quartile Discrepancy Rate
Description: Quartile discrepancies refer to the difference between
  the participant-recorded number of actuations and the participant-recorded
  counter readout at each of the 4 weekly visit intervals [ie, quartiles] to
  evaluate whether there was any difference in agreement over the life of
  the inhaler. The Quartile Discrepancy Rate was calculated as 100 multiplied by the total number of discrepancies per Quartile across all participant who used at least 90% of the labeled actuations divided by the total number of actuations per Quartile in the same population.
Time Frame: 4-week Treatment Period
Population: Completer Population, defined as participants who had recorded use of at least 90% of the labeled actuations during the 4-week Treatment Period.
Measure: Number; unit: discrepancies per 100 actuations
Arm/Group | MF/F MDI 100/10 mcg BID (With Dose Counter)
Number analyzed (Participants) | 233
discrepancies per 100 actuations | 0.13

3. Primary Outcome: Overall Discrepancy Size
Description: Discrepancy Size refers to the magnitude of the discrepancy between the dose counter readout and the number of recorded actuations (definition of discrepancy). Overall Discrepancy Size was calculated as 100 multiplied by the sum of the absolute values from each Dose Counter Discrepancy Size across all participants who used at least 90% of the labeled actuations divided by the total number of recorded actuations in the same participant population.
Time Frame: 4-week Treatment Period
Population: as for outcome 2
Measure: Number; unit: Discrepancy Size Per 100 actuations
Arm/Group | MF/F MDI 100/10 mcg BID (With Dose Counter)
Number analyzed (Participants) | 233
Discrepancy Size Per 100 actuations | 0.14

4. Primary Outcome: End of Use Agreement: Number of Inhalers With an End of Use Agreement of 0 (Completer Population)
Description: The difference in the final MDI dose counter readout and the total number of recorded actuations at the end-of-use. Dose Counter end-of-use agreement was calculated as the sum of the absolute difference between the final dose counter readout and the number of recorded actuations across all participants who used at least 90% of the labeled actuations (excluding participants who used the inhaler beyond the labeled number of actuations) divided by the total number of participants in this population. No participant used more than two inhalers during the treatment period.
Time Frame: 4-week Treatment Period
Population: Completer Population, excluding 2 participants who used more than the labeled number of actuations.
Measure: Number; unit: Number of inhalers
Arm/Group | MF/F MDI 100/10 mcg BID (With Dose Counter)
Number analyzed (Participants) | 233
Number of inhalers | 175

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Participants received open-label MF/F 100/10 mcg BID during the 2-week
  Screening Period and the 4-week Treatment Period. All participants who received at least one dose of MF/F were included in the safety analysis.
Groups:
- MF/F MDI 100/10 mcg BID: Included all participants that received 100/10 mcg BID (with and without dose counter)
Arm/Group | MF/F MDI 100/10 mcg BID
Serious Adverse Events (participants affected / at risk) | 1/272
Other Adverse Events (participants affected / at risk) | 0/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 100/10 mcg BID (N=272)
Oedema Peripheral (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish/present any interim results without prior sponsor written consent. The investigator agrees to provide to the sponsor, 45 days prior to submission, review copies for publication that report any study results. The sponsor has the right to review and comment. If the parties disagree, investigator agrees to meet with the sponsor, prior to submission for publication, to discuss and resolve any such issues/disagreement.